CLINICAL TRIAL: NCT01717924
Title: Multicenter Randomized Controlled Trial to Evaluate the Strategy of Primary Surgery Versus Primary Chemotherapy in Resectable Signet Ring Cell Gastric Adenocarcinoma (ADCI002 Study)
Brief Title: Evaluation of Surgery Versus Primary Chemotherapy in Resectable Signet Ring Cell Gastric Adenocarcinoma
Acronym: ADCI002
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other); UNICANCER (Other); Federation of Research in Surgery (FRENCH) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011_25; 2012-000998-24 (EudraCT Number)
Record Dates: First submitted 2012-10-23; First posted 2012-10-31 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Signet Ring Cell Gastric Adenocarcinoma
Keywords: Signet ring cell; gastric adenocarcinoma; peri-operative chemotherapy; surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- peri-operative chemotherapy (Active Comparator): Neoadjuvant chemotherapy with 3 cycles of Epirubicin/Cisplatin/5 fluoro-uracil (oral or intra-veinous) Surgery within 3 and 6 weeks after the end of neoadjuvant chemotherapy Adjuvant chemotherapy with 3 cycles of the same chemotherapy within 6 and 12 weeks after surgery
  Interventions: Procedure: peri-operative chemotherapy
- surgery first with adjuvant chemotherapy (Experimental): Surgery first Adjuvant chemotherapy with 3 cycles of Epirubicin/Cisplatin/5FU within 6 and 12 weeks after surgery No neoadjuvant chemotherapy
  Interventions: Procedure: Surgery first

INTERVENTIONS:
Procedure: peri-operative chemotherapy — Usual treatment strategy for gastric adenocarcinoma
  Arms: peri-operative chemotherapy
Procedure: Surgery first — strategy with a surgical procedure first, without the usual peri-operative chemotherapy
  Arms: surgery first with adjuvant chemotherapy

SUMMARY:
The ADCI 002 trial is a large multicenter phase II-III prospective randomized controlled trial comparing primary surgery versus primary chemotherapy followed by surgery in patients with a resectable signet ring cell gastric adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of the stomach or the oesogastric junction of type III of Siewert classification,histologically proven with the presence of signet ring cells (according to WHO 2000 classification) or diffuse form (according to Lauren classification) on pre-therapeutic biopsies
* tumoural stage IB, II or III (according to UICC-AJCC 2009)
* patient judged resectable in a curative intent on inclusion
* absence of distant metastasis
* absence of peritoneal carcinomatosis during pre-treatment explorative laparoscopy
* WHO performance status 2 or less
* age over 18 or under 80 years
* weight loss at the time of inclusion < 15%
* neutrophilic polynuclears more than 1500/mm3
* platelets more than 100000/mm3
* creatinine clearance more than 50 ml/min
* serum-albumin more than 30 gram/l
* bilirubin less than 1,5 normal
* prothrombin rate over 80%
* absence of prior treatment with chemotherapy or radiotherapy for gastric cancer
* absence of kniwn child B or C cirrhosis
* left ventricular ejection fraction more than 50% before epirubicin treatment
* extension check-up performed within 4 weeks of inclusion
* signed written informed consent given by the patient

Exclusion Criteria:

* no corresponding to the inclusion criteria
* another malignant tumour treated for curative purposes during the past 5 years excepted basocellular skin carcinoma or in situ uterine cervix cancer
* allergy to the active substance or one of the excipients in the study drugs
* pregnancy or breast-feeding
* any other concommitant treatment, immunotherapy or hormonal therapy
* history of abdominal or chest radiotherapy
* any evolving disorder which is not under control (liver failure, kidney failure, respiratory failure, evolving heart failure or myocardial necrosis during the past 6 months)
* patients who cannot be regularly monitored

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients dead in the 2-years | 2 years

SECONDARY OUTCOMES:
Disease-free survival at 2 years | 2 years
Disease-free survival at 3 years | 3 years
Overall survival at 3 years | 3 years
R0 resection rate | within 1 year
grade III/IV toxicity | 2 years
  tolerance will be measured by the rate and grade of chemotherapy's complications
post operative morbi-mortality | 2 years
Average of patients who benefit from the overall treatment strategy | 2 years
quality of life | 2 years
emotional status | 2 years
  It will be assessed by quality of life questionnaire(QLQ-C30, QLQ-STO-22,SF-36) and emotional status questionnaire(CES-D, STAI-Y-A, Brief-IPQ, WCC, ICEC-R, CRA)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume mariette, MD,PhD, Principal Investigator — FFCD, FNCLCC, FRENCH
Locations (1):
- General and digestive surgical department, Claude Huriez Hospital, University Hospital, Lille, France

REFERENCES:
- [Derived] Piessen G, Messager M, Le Malicot K, Robb WB, Di Fiore F, Guilbert M, Moreau M, Christophe V, Adenis A, Mariette C. Phase II/III multicentre randomised controlled trial evaluating a strategy of primary surgery and adjuvant chemotherapy versus peri-operative chemotherapy for resectable gastric signet ring cell adenocarcinomas - PRODIGE 19 - FFCD1103 - ADCI002. BMC Cancer. 2013 Jun 10;13:281. doi: 10.1186/1471-2407-13-281. PMID 23758655